CLINICAL TRIAL: NCT06258135
Title: At Home Placebo-controlled 8-week GOS Intervention on Emotion Behaviour and Cognition in Children (Age 6-14 Years).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FearlessStudy4
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Emotional Regulation
MeSH Terms: conditions — Emotional Regulation | interventions — 4'-galactooligosaccharide; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator)
  Interventions: Dietary Supplement: Galacto-oligosaccharide
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Galacto-oligosaccharide — Single 7g dose daily for 28 days
  Arms: Treatment
Dietary Supplement: Maltodextrin — Single 7g dose daily for 28 days
  Arms: Placebo

SUMMARY:
This study aims to investigate how GOS food supplement influences the gut-microbiome-brain axis to improve emotion regulation skills and cognition in a sample of children and adolescents (aged 6-14 years).

ELIGIBILITY:
Inclusion Criteria:

* Typically developing, healthy male or female aged 6-14 years
* Access to home laptop/ personal computer

Exclusion Criteria:

* Current clinical levels of anxiety and/or co-morbid psychological diagnoses
* Neuro/developmental disorders
* Gastro-intestinal problems or disease
* Restrictive diets (e.g., lactose intolerance, gluten free)

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in trait anxiety. | End of treatment (4 weeks), Follow up (8 weeks).
  Self report instrument: state-trait anxiety measure for children (STAIC) - Trait scale.
Changes in emotion processing. | End of treatment (4 weeks), Follow up (8 weeks).
  Performance on behavioural task: emotional dot-probe task.

SECONDARY OUTCOMES:
Changes in depression. | End of treatment (4 weeks), Follow up (8 weeks).
  Self report instrument: child depression inventory (CDI).
Changes in attention networks. | End of treatment (4 weeks), Follow up (8 weeks).
  Performance on behavioural task: attention network test (ANT) adapted for use by children.
Changes in nutrient intake | End of treatment (4 weeks), Follow up (8 weeks).
  Self report instrument: food diary completed over 4 days, average intakes calculated.

OTHER OUTCOMES:
Parental anxiety: covariate of child outcome. | Baseline, End of treatment (4 weeks), Follow up (8 weeks).
  Self report instrument: state-trait anxiety inventory (STAI) - Trait scale.
Parental emotion processing: covariate of child outcome. | Baseline, End of treatment (4 weeks), Follow up (8 weeks).
  Performance on behavioural task: emotional dot-probe task.
Parent depression | Baseline, End of treatment (4 weeks), Follow up (8 weeks).
  Self report instrument: Becks depression inventory (BDI-II).
Parent attention networks | Baseline, End of treatment (4 weeks), Follow up (8 weeks).
  Performance on behavioural task: attention network test.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnstone N, Cohen Kadosh K. Indicators of improved emotion behavior in 6-14-year-old children following a 4-week placebo controlled prebiotic supplement intervention at home with a parent. Nutr J. 2025 Mar 1;24(1):34. doi: 10.1186/s12937-025-01098-5. PMID 40025494